CLINICAL TRIAL: NCT00922636
Title: A Fixed-Dose, Randomized, Double-Blind, Placebo-Controlled Study of LY2216684 in Pediatric Patients With Attention Deficit/Hyperactivity Disorder
Brief Title: A Study of Pediatric Patients With Attention Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10925; H9P-MC-LNBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Methylphenidate; Tablets; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Methylphenidate (Active Comparator): Extended-release methylphenidate 18 milligrams per day (mg/day) to 54 mg/day, based on weight, given once daily (QD) and orally (po) as a capsule for the 8-week double-blind treatment phase, followed by 2 weeks of placebo in the taper phase.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (tablet); Drug: Placebo (capsule)
- LY2216684 (0.1 mg/kg/day) (Experimental): Taken in tablet form QD po for the 8-week double-blind treatment phase, followed by 2 weeks of placebo in the taper phase.
  Interventions: Drug: LY2216684
- LY2216684 (0.2 mg/kg/day) (Experimental): Taken in tablet form QD po for the 8-week double-blind treatment phase, followed by 2 weeks of tapering in the taper phase.
  Interventions: Drug: LY2216684
- LY2216684 (0.3 mg/kg/day) (Experimental): Taken in tablet form QD po for the 8-week double-blind treatment phase, followed by 2 weeks of tapering in the taper phase.
  Interventions: Drug: LY2216684

INTERVENTIONS:
Drug: LY2216684 — Taken in tablet form QD po.
  Other Names: Edivoxetine
  Arms: LY2216684 (0.1 mg/kg/day); LY2216684 (0.2 mg/kg/day); LY2216684 (0.3 mg/kg/day)
Drug: Methylphenidate — Extended-release methylphenidate 18 mg/day to 54 mg/day, based on weight, QD po as a capsule for the 8-week double-blind treatment phase.
  Arms: Methylphenidate
Drug: Placebo (tablet) — Placebo given as a tablet for LY2216684 blind QD po for the 8-week double-blind treatment phase, followed by 2 weeks in the taper phase.
  Arms: Placebo
Drug: Placebo (capsule) — Placebo given as a capsule for methylphenidate blind QD po for the 8-week double-blind treatment phase followed by 2 weeks in the taper phase.
  Arms: Placebo

SUMMARY:
The primary purpose of your child's participation in this study is to determine whether LY2216684 can help pediatric patients with attention-deficit/hyperactivity disorder (ADHD); and assess the safety of LY2216684 and any side effects that might be associated with it.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnostic criteria for ADHD based on Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime (K-SADS-PL) prior to randomization.
* Patients must have an Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHD-RS-IV-PV:IR) total score at least 1.5 standard deviations above the age/gender norm prior to randomization. They must have a Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) score greater than or equal to 4 at both the patients screening visit, prior to randomization.
* Patients must have laboratory results; showing no clinically significant abnormalities.
* Patients must be of normal intelligence, as assessed by the investigator.
* Patients/parents must have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including venous punctures and examinations required by the protocol.
* Patients of child-bearing potential agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug. Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment based on a urine pregnancy test.

Exclusion Criteria:

* Patients who weigh less than 18 kg or greater than 75 kg at screening and at randomization.
* Female patients who are pregnant or who are breast-feeding. Patients who have a history of Bipolar I/ II, psychosis, or pervasive developmental disorder.
* Patients who have current motor tics or a diagnosis of Tourette's Syndrome.
* Patients with marked anxiety, tension, and agitation sufficient, to contraindicate treatment with extended-release methylphenidate.
* Patients with a history of any seizure disorder, known electroencephalographic (EEG) abnormalities in the absence of seizures.
* If the electrocardiogram (ECG) assessed at screening/prior to randomization shows an abnormality meeting one or more of the absolute exclusion criteria listed in the Pediatric ECG Alert Criteria must be excluded from the study.
* Patients who, in the opinion of the investigator, are at serious suicidal risk.
* Patients with a history of severe allergies to more than one class of medications, multiple adverse drug reactions, or known hypersensitivity to extended-release methylphenidate.
* Patients with a history of alcohol or drug abuse within the past 3 months prior to, or who are currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner that the investigator considers indicative of abuse.
* Patients who screen positive for drugs of abuse not prescribed by a physician cannot participate. Drug screen may be repeated at the discretion of the investigator, and the patient may be allowed to enter the study if the repeat screen is negative. All patients must have a negative drug screen before enrollment in the study.
* Patients who have a medical condition that would increase sympathetic nervous system activity markedly, or who are taking a medication on a daily basis that has sympathomimetic activity are excluded. Such medications can be taken on an as-needed basis.
* Patients with problems that would be exacerbated by increased norepinephrine tone, including a history of cardiovascular disease, thyroid dysfunction, glaucoma, urinary retention, or severe gastrointestinal narrowing.
* Patients who, at any time during the study, are likely to need psychotropic medications apart from the drugs under study.
* Patients who, at any time during the study, are likely to begin structured psychotherapy aimed at ADHD symptoms are excluded. Psychotherapy initiated at least 1 month prior to screening is acceptable.
* Patients who have used a monoamine oxidase inhibitor (MAOI) during the 2 weeks prior to randomization.
* Patients with current or past history of clinically significant hypertension.
* Patients who are currently enrolled in, or discontinued within the last 30 days from a clinical trial involving an off-label use of an investigational drug, or concurrently enrolled in any other type of medical research.
* Patients who have participated in a prior study of LY2216684.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norristown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wharton, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce, Puerto Rico

REFERENCES:
- [Derived] Lin DY, Kratochvil CJ, Xu W, Jin L, D'Souza DN, Kielbasa W, Allen AJ. A randomized trial of edivoxetine in pediatric patients with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2014 May;24(4):190-200. doi: 10.1089/cap.2013.0043. PMID 24840045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment phase: Participants were randomized to:
  1 of 3 fixed-dose LY2216684 treatment arms, placebo, or extended-release methylphenidate (stimulant-naive stratum)
  1 of 3 fixed-dose LY2216684 treatment arms or placebo only (stimulant-prior stratum) Optional Taper phase: Participants received study drug (at reduced dose) or placebo for 2 weeks
Groups:
- Methylphenidate: Participants were given 18 milligrams per day (mg/day) to 54 mg/day of extended-release methylphenidate capsules, based on weight, once daily (QD) and orally (po) for the 8-week double-blind treatment phase, followed by 2 weeks of placebo in the optional taper phase. Participants were also given placebo tablets to maintain LY2216684 blinding during the double-blind treatment phase.
- Placebo: Participants were given the placebo in both tablet (LY2216684 placebo) and capsule (methylphenidate placebo) forms QD po for the 8-week double-blind treatment phase, followed by 2 weeks of placebo in the optional taper phase.
- LY2216684 (0.1 mg/kg/Day): Participants were given 0.1 mg/kg/day of LY2216684 in tablet form QD po for the 8-week double-blind treatment phase, followed by 2 weeks of placebo in the optional taper phase. Participants were also given placebo capsules to maintain methylphenidate blinding.
- LY2216684 (0.2 mg/kg/Day): Participants were given 0.2 mg/kg/day of LY2216684 in tablet form QD po for the 8-week double-blind treatment phase, followed by 2 weeks of tapering in optional taper phase. Participants were also given placebo capsules to maintain methylphenidate blinding.
- LY2216684 (0.3 mg/kg/Day): Participants were given 0.3 mg/kg/day of LY2216684 in tablet form QD po for the 8-week double-blind treatment phase, followed by 2 weeks of tapering in the optional taper phase. Participants were also given placebo capsules to maintain methylphenidate blinding.
Period: Overall Study
Arm/Group | Methylphenidate | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Started | 36 | 78 | 76 | 75 | 75
Entered Optional Taper Phase | 4 | 10 | 15 | 7 | 12
Completed | 29 | 62 | 56 | 58 | 59
Not Completed | 7 | 16 | 20 | 17 | 16
Not completed — Adverse Event | 3 | 3 | 2 | 3 | 2
Not completed — Lack of Efficacy | 1 | 7 | 3 | 2 | 4
Not completed — Sponsor Decision | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 2 | 2 | 0
Not completed — Entry Criteria Not Met | 0 | 0 | 1 | 1 | 0
Not completed — Parent/Caregiver Decision | 2 | 4 | 3 | 5 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day) | Total
Number analyzed (Participants) | 36 | 78 | 76 | 75 | 75 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.92 (2.94) | 11.37 (3.07) | 11.90 (3.03) | 12.59 (2.81) | 11.47 (3.10) | 11.63 (3.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 25 | 24 | 22 | 20 | 100
  Male | 27 | 53 | 52 | 53 | 55 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 20 | 21 | 20 | 19 | 89
  Not Hispanic or Latino | 27 | 58 | 55 | 55 | 56 | 251
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 1 | 1 | 4
  Asian | 0 | 4 | 5 | 3 | 5 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 8 | 9 | 10 | 12 | 45
  White | 25 | 60 | 55 | 57 | 50 | 247
  More than one race | 5 | 6 | 5 | 4 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 4 | 4 | 5 | 4 | 18
  Mexico | 0 | 0 | 1 | 0 | 1 | 2
  Puerto Rico | 2 | 3 | 4 | 2 | 3 | 14
  Taiwan | 0 | 4 | 5 | 3 | 4 | 16
  United States | 33 | 67 | 62 | 65 | 63 | 290

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHD-RS-IV-PV:IR) Total Score at Week 8
Description: Assesses 18 Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision ADHD diagnosis symptoms/severity in past week. Each item: 0 (none/never, rarely) to 3 (severe/very often). Total score ranges from 0 to 54. Higher total scores indicate greater illness severity. Change scores=Week 8 score-baseline score. Least Squares (LS) Mean Change adjusted for fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: Per protocol (PP) population included all randomized participants with a baseline and at least 1 post-baseline result, excluding data from participants whose data might have been compromised.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 58 | 60 | 59
units on a scale | -10.35 (1.52) | -12.20 (1.63) | -16.09 (1.53) | -16.39 (1.57)
Statistical Analysis 1: Comparison: Placebo vs LY2216684 (0.2 mg/kg/Day); Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — Statistical significance was assessed at an alpha level of 0.027 with a Dunnett adjustment for multiple comparisons; The Least Squares (LS) Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis; Mean Difference (Final Values) = -5.74 — The LS Mean difference was computed as treatment minus placebo
Statistical Analysis 2: Comparison: Placebo vs LY2216684 (0.3 mg/kg/Day); Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — Statistical significance was assessed at an alpha level of 0.027 with a Dunnett adjustment for multiple comparisons; The Least Squares (LS) Mean Value is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis; Mean Difference (Final Values) = -6.04 — The LS Mean difference was computed as treatment minus placebo

2. Secondary Outcome: Change From Baseline in the Swanson, Nolan and Pelham Questionnaire: Attention-Deficit/Hyperactivity Disorder Subscale (SNAP-IV: ADHD) Total Score at Week 8
Description: Includes Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision ADHD criteria for inattention (items 1-9) and hyperactivity/impulsivity (items 11-19) symptom subsets. Item score: 0 (not at all) to 3 (very much) rating scale. Total score is average of 18 items. Higher total scores=greater ADHD symptoms. Least Squares Mean change is adjusted for fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and the continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: Per protocol (PP) participant population included all randomized participants with a baseline and at least 1 post-baseline result, excluding data from participants whose data may have been compromised.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 13 | 9 | 7 | 10
units on a scale | 0.10 (0.25) | 0.35 (0.26) | -0.21 (0.24) | -0.46 (0.20)

3. Secondary Outcome: Change From Baseline in the Swanson, Nolan and Pelham Questionnaire: Attention-Deficit/Hyperactivity Disorder Subscale (SNAP-IV: ADHD) Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 2
Time Frame: Baseline, 8 weeks
Population: Stimulant naive participants randomized to methylphenidate with a baseline and at least 1 post-baseline result but excluded the participants whose data may have been compromised.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 3
units on a scale | NA (NA) — Sample size not able to be analyzed.

4. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS) Academic Difficulties Total Score and the Language and Math Subscales at Week 8
Description: The CP-CBRS academic difficulties total/language/math subscale score is a measure of academic performance. Each subscale item score ranges from 0 (never, seldom) to 3 (very often, very frequently). Total score is expressed as T-score based on gender/age norms. Academic difficulties T-score range: 0-100. Higher T-scores denote greater academic difficulties. Change scores=Week 8 score-baseline score. Least Squares Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis adjusted for fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline total score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: Per protocol (PP) population included all randomized participants with a baseline and at least 1 post-baseline result, excluding data from participants whose data may have been compromised.
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score
  Total Score | -6.09 (1.43) | -6.13 (1.53) | -5.93 (1.46) | -12.53 (1.49)
  Language Subscale Score | -5.87 (1.43) | -6.75 (1.54) | -6.07 (1.45) | -12.5 (1.49)
  Math Subscales Score | -4.63 (1.67) | -3.8 (1.79) | -2.85 (1.7) | -7.78 (1.74)
Statistical Analysis 1: Comparison: Placebo vs LY2216684 (0.2 mg/kg/Day); Gated secondary analysis for total score. If both LY2216684 groups (0.2 mg/kg/day and 0.3 mg/kg/day) were statistically significantly superior than placebo for the primary endpoint, then gated secondary analysis was assessed at an alpha level of 0.027. If only 0.2 mg/kg/day or 0.3 mg/kg/day LY2216684 was statistically significantly superior than placebo for the primary endpoint, then gated secondary analysis was assessed at an alpha level of 0.023 for the corresponding group; Test type: Superiority or Other; p = 0.938, Mixed Models Analysis — Statistical significance was assessed at an alpha level of 0.027 with a Dunnett adjustment for multiple comparisons; Least squares (LS) mean is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis; Mean Difference (Final Values) = 0.16
Statistical Analysis 2: Comparison: Placebo vs LY2216684 (0.3 mg/kg/Day); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Statistical significance was assessed at an alpha level of 0.027 with a Dunnett adjustment for multiple comparisons; Least squares (LS) mean is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis; Mean Difference (Final Values) = -6.44

5. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS) Academic Difficulties Total Score and the Language and Math Subscales at Week 8 in Stimulant Naive Methylphenidate Group
Description: The CP-CBRS academic difficulties total/language/math subscale score is a measure of academic performance. Each subscale item score ranges from 0 (never, seldom) to 3 (very often, very frequently). Total score is expressed as T-score based on gender/age norms. Academic difficulties T-score range: 0-100. Higher T-scores denote greater academic difficulties. Change scores=Week 8 score-baseline score. Least Squares Mean Change is adjusted for fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline total score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score
  Total Score | -12.14 (2.30)
  Language Subscale Score | -12.24 (2.32)
  Math Subscales Score | -7.11 (2.68)

6. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) Total Score at Week 8
Description: Measures participant's overall ADHD symptom severity. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Higher scores represent greater illness severity. Change scores=Week 8 score-baseline score. The Least Squares (LS) Mean Change was based on the fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, as well as the continuous, fixed effects of baseline CGI-S score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 62 | 59 | 60 | 59
units on a scale | -1.07 (0.15) | -0.96 (0.16) | -1.52 (0.15) | -1.41 (0.16)

7. Secondary Outcome: Change From Baseline in the Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 6
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 26
units on a scale | -1.69 (0.25)

8. Secondary Outcome: Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Improvement Scale (CGI-ADHD-I) Endpoint Score During the Treatment Phase (Weeks 1-8)
Description: Measures total improvement (or worsening) of a participant's ADHD symptoms from the beginning of treatment. Scores range from 1 (very much improved) to 7 (very much worsened). Lower scores represent greater improvement. Least Squares (LS) Mean Change for weeks 1-8 is from a restricted maximum likelihood-based, mixed model repeated measure analysis. The model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction.
Time Frame: Weeks 1 through 8
Population: Per protocol (PP) population included all randomized participants with a post-baseline result, excluding data from participants whose data may have been compromised.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 59 | 60 | 59
units on a scale | 3.05 (0.14) | 3.01 (0.15) | 2.54 (0.14) | 2.53 (0.15)

9. Secondary Outcome: Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Improvement Scale (CGI-ADHD-I) Endpoint Score During the Treatment Phase (Weeks 1-8) in Stimulant Naive Methylphenidate Group
Description: as for outcome 8
Time Frame: Weeks 1 through 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Total Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 26
Total Score | 2.31 (0.23)

10. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR ADHD) Predominantly Hyperactive-Impulsive Type and Predominantly Inattentive Type Total Score and Symptom Scores at Week 8
Description: Measures ADHD symptom severity. Individual items on each subscale are scored from 0 (never) to 3 (very often). Total score expressed as T-score based on gender/age norms. Subscale total T-scores (0-100); higher T-scores=greater symptom severity. Least Squares Mean Change is from restricted maximum likelihood-based, mixed model repeated measure analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline total score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score
  Predominantly Hyperactive-Impulsive Type Total | -8.70 (1.71) | -6.30 (1.84) | -12.94 (1.75) | -15.69 (1.78)
  Predominantly Inattentive Type Total Scale | -10.71 (1.62) | -8.32 (1.74) | -10.99 (1.66) | -16.99 (1.69)

11. Secondary Outcome: Change From Baseline in the CP-CBRS DSM-IV-TR ADHD Predominantly Hyperactive-Impulsive Type and Predominantly Inattentive Type Total Score and Symptom Scores at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 10
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score
  Predominantly Hyperactive-Impulsive Type Total | -12.41 (2.64)
  Predominantly Inattentive Type Total Scale | -18.28 (2.63)

12. Secondary Outcome: Change From Baseline in the Swanson, Nolan and Pelham (SNAP-IV) Oppositional Defiant Disorder (ODD) Total Score at Week 8
Description: Measures oppositional defiance disorder symptoms. Total scores range from 0 (not at all) to 3 (very much). Higher total scores represent greater ODD. Change scores=Week 8 score-baseline score. Least Squares Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline total score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 13 | 9 | 7 | 11
units on a scale | 0.19 (0.16) | 0.62 (0.18) | -0.04 (0.17) | -0.30 (0.13)

13. Secondary Outcome: Change From Baseline in the Swanson, Nolan and Pelham (SNAP-IV) Oppositional Defiant Disorder (ODD) Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 12
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 3
units on a scale | -0.72 (0.38)

14. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS) Impairment Items Subscales-Total Score at Week 8
Description: Rates schoolwork/grades, friendships/relationships, home life functioning (0=never to 3=very often). Total score expressed as a T-score based on gender/age norms (range 0-100). Higher T-score=greater symptom severity. Change scores=Week 8 score-baseline score. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis; included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score
  Schoolwork/Grades Score | -0.49 (0.12) | -0.35 (0.13) | -0.53 (0.12) | -0.81 (0.13)
  Friendships/Relationships Score | -0.43 (0.12) | -0.00 (0.13) | -0.22 (0.12) | -0.65 (0.13)
  Home Life Score | -0.40 (0.12) | -0.08 (0.13) | -0.44 (0.13) | -0.73 (0.13)

15. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS) Impairment Items Subscales-Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 14
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score
  Schoolwork/Grades Score | -0.65 (0.19)
  Friendships/Relationships Score | -0.28 (0.20)
  Home Life Score | -0.44 (0.21)

16. Secondary Outcome: Number of Participants With Suicidal Behaviors, Ideations, and Acts Based on The Columbia Suicide Severity Rating Scale (C-SSRS) at Week 8
Description: Captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors, ideations, and acts are provided. Suicidal behavior: a "yes" answer to any of 3 suicidal behavior questions: preparatory acts or behavior, aborted attempt, and interrupted attempt. Suicidal ideation: "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation. Suicidal act: a "yes" answer to actual attempt or completed suicide, nonfatal suicide attempt, and completed suicide.
Time Frame: 8 weeks
Population: Intent to treat (ITT). All randomized participants with a baseline and at least 1 post-baseline C-SSRS assessment.
Measure: Number; unit: Participants
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 78 | 75 | 73 | 73
Participants
  Suicidal Ideation | 1 | 1 | 5 | 2
  Suicidal Behavior | 0 | 0 | 0 | 0
  Suicidal Acts | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Suicidal Behaviors, Ideations, and Acts Based on The Columbia Suicide Severity Rating Scale (C-SSRS) at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 16
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Methylphenidate
Number analyzed (Participants) | 35
Participants
  Suicidal Ideation | 1
  Suicidal Behavior | 0
  Suicidal Acts | 0

18. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Symptom Subscale for Manic Episode - Total Score at Week 8
Description: Measures manic symptom severity. Individual subscale items range: 0 (never) to 3 (very often). Total score expressed as T-score based on gender/age norms (0-100). Higher T-scores=greater symptom severity. Change scores=Week 8 score-baseline score. Least Squares Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 56
T-Score | -9.35 (1.74) | -5.00 (1.88) | -12.60 (1.79) | -12.41 (1.85)

19. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Symptom Subscale for Manic Episode - Total Score at 8 Weeks in Stimulant Naive Methylphenidate Group
Description: as for outcome 18
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score | -11.85 (2.76)

20. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS) Content Subscales - Total Score at Week 8
Description: Assess aggressive behaviors, academic difficulties, social problems, violence potential. Individual subscale items range: 0=never to 3=very often. Total expressed as T-score based on gender/age norms (0-100). Change scores=Week 8 score-baseline score. Least Squares (LS) Mean Change from restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis; included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score, baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score
  Aggressive Behaviors Scale Score | -5.52 (1.55) | -3.32 (1.68) | -8.09 (1.59) | -11.01 (1.62)
  Social Problems T-score | -6.77 (1.52) | -3.33 (1.63) | -5.19 (1.55) | -12.06 (1.58)
  Violence Potential T-score | -6.97 (1.36) | -4.22 (1.46) | -7.95 (1.39) | -11.88 (1.42)

21. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS) Content Subscales - Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 20
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score
  Aggressive Behaviors Scale Score | -10.96 (2.43)
  Social Problems T-score | -2.12 (2.50)
  Violence Potential T-score | -9.58 (2.11)

22. Secondary Outcome: Change From Baseline in the Child Health and Illness Profile-Adolescent Edition (CHIP-AE) Domain Scores at Week 8
Description: Assesses adolescent's health status/functioning level. Domains: Achievement, Satisfaction, Comfort, Risk Avoidance, Resilience. Items assess frequency of activities/feelings (1=never, 5=always). Standard scores (T-scores) calculated for all domains by adjusting raw scores based on established reference group mean, standard deviation (T-scores mean=50, standard deviation=10). Higher scores=better health. Least Squares (LS) Mean Change from analysis of covariance model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), and baseline score.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 30 | 32 | 32 | 26
T-Score
  Achievement Section (n=3,3,4,3) | -339.71 (0.00) | 301.79 (0.00) | -12.42 (0.00) | 64.55 (0.00)
  Discomfort Section (n=30,31,32,26) | -1.29 (1.03) | 0.99 (1.07) | 1.10 (0.98) | 2.39 (1.14)
  Resilience Section (n=30,30,31,26) | 1.90 (1.38) | 0.21 (1.45) | 1.62 (1.33) | 1.28 (1.49)
  Risks Section (n=30,30,31,26) | -0.08 (1.20) | -0.28 (1.27) | 2.18 (1.16) | 0.74 (1.32)
  Satisfaction Section (n=30,32,32,26) | -0.12 (1.43) | -0.05 (1.44) | 2.95 (1.35) | 0.72 (1.55)

23. Secondary Outcome: Change From Baseline in the Child Health and Illness Profile-Adolescent Edition (CHIP-AE) Domain Scores at Week 8 in Stimulant Naive Methylphenidate Group
Description: Assesses adolescent's health status/functioning level. Domains: Achievement, Satisfaction, Comfort, Risk Avoidance, Resilience. Items assess frequency of activities/feelings (1=never, 5=always). Standard scores (T-scores) calculated for all domains by adjusting raw scores based on established reference group mean, standard deviation (T-scores mean=50, standard deviation=10). Higher scores=better health. Least squares (LS) mean of the change from baseline to endpoint (week 8) is from an ANCOVA model. The model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), and baseline CHIP-AE domain score.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 6
T-Score
  Achievement Section (n=1) | NA (NA) — Sample size not able to be analyzed.
  Discomfort Section (n=6) | -1.97 (2.47)
  Resilience Section (n=6) | -4.06 (3.21)
  Risks Section (n=6) | 2.01 (3.06)
  Satisfaction Section (n=6) | 2.19 (3.25)

24. Secondary Outcome: Change From Baseline in the Child Health and Illness Profile - Child Edition (CHIP-CE) at Week 8
Description: 76-item parent-rated assessment of child's health status/functioning level. Most items assess frequency of activities/feelings (1=never, 5=always). Standard scores (T-scores) were calculated for all domains by adjusting raw scores based on an established reference group mean and standard deviation (T-scores mean=50, standard deviation=10). Higher scores denote improvement. Least Squares (LS) Mean Change is from an analysis of covariance model that included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), and baseline domain score.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 28 | 16 | 19 | 29
T-Score
  Achievement Standardized Score (n=27,14,19,26) | 3.82 (1.65) | 3.45 (2.48) | 2.96 (2.08) | 3.81 (1.70)
  Comfort Standardized Score (n=28,16,19,29) | 8.24 (1.69) | 2.96 (2.45) | 3.50 (2.17) | 7.82 (1.72)
  Resilience Standardized Score (n=28,16,19,29) | 4.07 (1.96) | 0.60 (2.82) | 0.19 (2.53) | 4.75 (1.98)
  Risk Avoidance Standardized Score (n=28,16,19,29) | 6.06 (1.73) | 1.81 (2.57) | 5.77 (2.20) | 4.75 (1.74)
  Satisfaction Standardized Score(n=28,16,19,29) | 1.19 (1.72) | -2.07 (2.50) | -1.24 (2.27) | 3.63 (1.72)

25. Secondary Outcome: Change From Baseline in the Child Health and Illness Profile - Child Edition (CHIP-CE) at Week 8 in Stimulant Naive Methylphenidate Group
Description: 76-item parent-rated assessment of child's health status/functioning level. Most items assess frequency of activities/feelings (1=never, 5=always). Standard scores (T-scores) were calculated for all domains by adjusting raw scores based on an established reference group mean and standard deviation (T-scores mean=50, standard deviation=10). Higher scores denote improvement. Least Squares (LS) Mean Change is from an analysis of ANCOVA model that included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), and baseline domain score.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 18
T-Score
  Achievement Standardized Score (n=17) | 5.21 (2.02)
  Comfort Standardized Score (n=18) | 4.06 (1.93)
  Resilience Standardized Score (n=18) | 5.10 (2.62)
  Risk Avoidance Standardized Score (n=18) | 6.97 (2.11)
  Satisfaction Standardized Score(n=18) | 1.90 (2.40)

26. Secondary Outcome: Change From Baseline in the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) Letter-Number Sequencing Score at Week 8
Description: Working memory subtest. Task involves sequencing, mental manipulation, attention, short-term memory, visual spatial imaging, and processing speed; consists of 10 items, 3 trials each. Scaled scores range: 1 to 19. Higher scores denote better performance. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis that included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 56 | 50 | 55 | 51
units on a scale | 1.30 (0.31) | 1.36 (0.33) | 1.48 (0.32) | 1.84 (0.33)

27. Secondary Outcome: Change From Baseline in the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) Letter-Number Sequencing Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 26
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 23
units on a scale | 1.58 (0.50)

28. Primary Outcome: Change From Baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHD-RS-IV-PV:IR) Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: Assesses 18 Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision ADHD diagnosis symptoms/severity in past week. Each item: 0 (none/never, rarely) to 3 (severe/very often). Total score ranges from 0 to 54. Higher total scores indicate greater illness severity. Change scores=Week 8 score-baseline score. LS Mean Change adjusted for fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 26
units on a scale | -19.46 (2.50)

29. Secondary Outcome: Change From Baseline in the Rapid Automatized Naming/Rapid Alternating Stimulus Test (RAN/RAS) Subtotal Scores at Week 8
Description: Assesses ability to accurately and rapidly recognize and name visual symbols. The tests consist of rapid automatized naming tests (that is, Letters, Numbers, Objects, Colors) and 2 rapid alternating stimulus tests (that is, 2-Set Letters and Numbers; 3-Set Letters, Numbers, and Colors). Scores are based on the amount of time required to name all the stimulus items in each test section. Raw scores were converted to standard scores based on participant's age and conversion tables from manual (mean=100, standard deviation=15). Higher scores=better ability. Least Squares (LS) Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 28 | 26 | 30 | 23
units on a scale
  Objects (n=21,18,18,11) | -0.56 (2.35) | 6.45 (2.42) | 11.70 (2.59) | 5.64 (3.61)
  Colors (n=25, 21, 26, 16) | 2.85 (1.76) | 4.86 (1.99) | 3.30 (1.82) | 2.98 (2.25)
  Numbers (n=28, 26, 30, 23) | 3.44 (1.14) | 2.85 (1.25) | 2.99 (1.09) | 2.38 (1.26)
  Letters (n=27,24,27,22) | 1.16 (1.37) | 2.84 (1.57) | 3.62 (1.57) | 2.22 (1.80)
  2-set Letters and Numbers (n=27, 23, 28, 19) | 5.23 (1.58) | 3.21 (1.60) | 6.38 (1.61) | 4.69 (1.91)
  3-set Letters, Numbers, and Colors (n=26,24,28,21) | 7.89 (1.90) | 3.86 (1.92) | 6.47 (1.82) | 1.56 (2.18)

30. Secondary Outcome: Change From Baseline in the Rapid Automatized Naming/Rapid Alternating Stimulus Test (RAN/RAS) Subtotal Scores at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 29
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 14
units on a scale
  Objects (n=9) | 0.65 (4.88)
  Colors (n=11) | 3.37 (2.94)
  Numbers (n=14) | 6.60 (2.16)
  Letters (n=11) | 7.81 (2.70)
  2-set Letters and Numbers (n=12) | 6.65 (2.57)
  3-set Letters, Numbers, and Colors (n=12) | 4.82 (2.91)

31. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Symptom Subscale for Oppositional Defiant Disorder (ODD) Total Score at Week 8
Description: Assess ODD symptom severity. Individual subscale items range from 0 (never) to 3 (very often/frequently). Total is expressed as a T-score based on gender/age norms (range 0-100). Higher T-score=greater ODD. Change scores=Week 8 score-baseline score. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: Per protocol (PP) population included all randomized participants with a baseline at least 1 post-baseline result, excluding data from participants whose data may have been compromised.
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score | -7.17 (1.52) | -4.00 (1.64) | -10.18 (1.57) | -12.29 (1.59)

32. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Symptom Subscale for Oppositional Defiant Disorder (ODD) Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 31
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score | -13.83 (2.54)

33. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Generalized Anxiety Disorder (GAD) and Separation Anxiety Disorder Symptom Subscales at Week 8
Description: Assess anxiety symptom severity. Individual subscale items: 0 (never, seldom) - 3 (very often/frequently). Total score expressed as T-score based on gender/age norms (0-100). Higher T-scores=greater anxiety. Change scores=Week 8 score-baseline score. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score
  CBRS Generalized Anxiety Disorder T-score | -9.09 (1.46) | -5.34 (1.57) | -11.07 (1.50) | -15.39 (1.53)
  CBRS Separation Anxiety Disorder Scale T-score | -6.71 (1.48) | -1.13 (1.59) | -5.88 (1.52) | -8.60 (1.54)

34. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Generalized Anxiety Disorder (GAD) and Separation Anxiety Disorder Symptom Subscales at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 33
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score
  CBRS Generalized Anxiety Disorder T-score | -8.78 (2.40)
  CBRS Separation Anxiety Disorder Scale T-score | -2.91 (2.66)

35. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Conduct Disorder Symptom Subscale Score at Week 8
Description: Assess conduct disorder symptom severity. Individual subscale items: 0 (never/seldom) - 3 (very often/frequently). Total expressed as T-score based on gender/age norms (0-100). Higher T-score=greater conduct disorder. Change scores=Week 8 score-baseline score. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis; included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score | -4.64 (1.43) | -2.24 (1.55) | -6.26 (1.48) | -7.62 (1.50)

36. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Conduct Disorder Symptom Subscale Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 35
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score | -7.10 (2.27)

37. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Major Depressive Episode Score at Week 8
Description: Assess depressive symptom severity. Individual subscale items range: 0 (never, seldom) to 3 (very often/frequently). Total expressed as T-score based on gender/age norms (0-100). Higher T-scores=greater depression. Change scores=Week 8 score-baseline score. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis and included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 60 | 52 | 58 | 57
T-Score | -10.27 (1.56) | -5.41 (1.68) | -9.58 (1.59) | -13.67 (1.62)

38. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Major Depressive Episode Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 37
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
T-Score | -1.09 (2.38)

39. Secondary Outcome: Change From Baseline in the Weekly Parent Ratings of Evening and Morning Behavior-Revised (WPREMB-R) Total Score at Week 8
Description: Parent-completed 11-item questionnaire (3 morning items, 8 evening items) on a scale of 0 (no difficulty) to 3 (a lot of difficulty). Total score ranges from 0 to 33; higher score=greater difficulty in evening and morning behavior. Least Squares (LS) Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis and includes fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 58 | 59 | 57
units on a scale | -4.95 (0.83) | -4.72 (0.89) | -7.08 (0.84) | -8.24 (0.87)

40. Secondary Outcome: Change From Baseline in the Weekly Parent Ratings of Evening and Morning Behavior-Revised (WPREMB-R) Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 39
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 25
units on a scale | -6.88 (1.45)

41. Secondary Outcome: Change From Baseline in the Weekly Parent Ratings of Evening and Morning Behavior-Revised (WPREMB-R) Morning Summary Score at Week 8
Description: Measures difficulty level of 3 common morning behaviors (for example, get out of bed) from 0 (no difficulty) to 3 (a lot of difficulty). Total score range is from 0 to 9; a higher score indicates greater difficulty in morning behavior. Least Squares (LS) Mean Change from restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis and includes fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline morning score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 58 | 59 | 58
units on a scale | -1.07 (0.28) | -0.91 (0.30) | -1.53 (0.29) | -2.20 (0.29)

42. Secondary Outcome: Change From Baseline in the Weekly Parent Ratings of Evening and Morning Behavior-Revised (WPREMB-R) Morning Summary Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 41
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 26
units on a scale | -0.80 (0.44)

43. Secondary Outcome: Change From Baseline in the Weekly Parent Ratings of Evening and Morning Behavior-Revised (WPREMB-R ) Evening Summary Score at Week 8
Description: Measures difficulty level of 8 common evening behaviors (for example, sit through dinner) from 0 (no difficulty) to 3 (a lot of difficulty). Total score ranges: 0 to 24; higher scores indicate greater difficulty in evening behavior. Least Squares (LS) Mean Change is from restricted maximum likelihood-based, mixed model repeated measure analysis (MMRM) and included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline evening score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 58 | 60 | 58
units on a scale | -3.34 (0.58) | -3.37 (0.61) | -4.77 (0.58) | -5.24 (0.60)

44. Secondary Outcome: Change From Baseline in the Weekly Parent Ratings of Evening and Morning Behavior-Revised (WPREMB-R ) Evening Summary Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 43
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 25
units on a scale | -6.17 (1.04)

45. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Mixed Episode Score at Week 8
Description: The mixed episode score does not exist in the Conners CBRS scale; therefore no analyses could be conducted.
Time Frame: Baseline, 8 weeks
Population: No participants had data analyzed because the mixed episode score does not exist in the outcome measure; therefore, no analyses could be conducted.
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 0 | 0 | 0 | 0

46. Secondary Outcome: Change From Baseline in the Conners' Comprehensive Behavior Rating Scale (CP-CBRS DSM-IV-TR) Mixed Episode Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: The mixed episode score does not exist in the Conners CBRS scale; therefore no analyses could be conducted.
Time Frame: Baseline, 8 weeks
Population: as for outcome 45
Arm/Group | Methylphenidate
Number analyzed (Participants) | 0

47. Secondary Outcome: Change From Baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Hyperactivity-Impulsivity and Inattention Subtotal Scores at Week 8
Description: Measures ADHD diagnostic symptoms (0=none/never-3=severe/very often). Inattention=sum odd items; hyperactivity-impulsivity=sum even items (subtotal: 0-27). Total scores: 0-54. High score=greater illness severity. Missing data-imputation in manual was applied. Least Squares Mean Change from restricted maximum likelihood-based, mixed model repeated measure analysis; included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 59 | 60 | 59
units on a scale
  Hyperactivity-Impulsivity Score (n=63, 58,60,59) | -4.88 (0.79) | -5.94 (0.84) | -7.53 (0.80) | -7.32 (0.81)
  Inattention Score (n=63, 59, 60, 59) | -5.55 (0.92) | -6.23 (0.98) | -8.58 (0.92) | -9.09 (0.94)

48. Secondary Outcome: Change From Baseline in the ADHDRS-IV-Parent:Inv Hyperactivity-Impulsivity and Inattention Subtotal Scores at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 47
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 26
units on a scale
  Hyperactivity-Impulsivity Score | -9.00 (1.29)
  Inattention Score | -10.46 (1.46)

49. Secondary Outcome: Change From Baseline in the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) Digit Span Total Score at Week 8
Description: A working memory subtest of WISC-IV, a measure of attention; concentration; sequencing; number facility; and auditory short-term memory. Scaled scores range from 1 to 19. Higher scores denote better performance. Least Squares (LS) Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure (MMRM) analysis and included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, as well as the continuous, fixed effects of baseline Digit Span total score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 56 | 51 | 56 | 51
units on a scale | 0.64 (0.30) | 1.22 (0.32) | 0.95 (0.30) | 1.02 (0.32)

50. Secondary Outcome: Change From Baseline in the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) Digit Span Total Score at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 49
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
units on a scale | 0.54 (0.47)

51. Secondary Outcome: Change From Baseline in the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) Digit Span Subtotal Scores at Week 8
Description: Measures attention, concentration, sequencing, number facility, and auditory short-term memory. Digit forward and digit backward subscales each comprise 2 trials and 8 items. Scaled scores range from 1 to 19. Higher scores denote better performance. Least Squares Mean Change is from a restricted maximum likelihood-based, mixed model repeated measure analysis. Model included fixed class effects of treatment, pooled investigative site, strata (prior stimulant use status), visit, and treatment*visit interaction, and continuous, fixed effects of baseline score and baseline score*visit interaction.
Time Frame: Baseline, 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 56 | 51 | 56 | 51
units on a scale
  Digit Span Forward: Scaled Process Score | 0.43 (0.31) | 0.97 (0.33) | 0.56 (0.31) | 0.61 (0.33)
  Digit Span Backward: Scaled Process Score | 0.77 (0.34) | 0.98 (0.37) | 1.04 (0.35) | 0.74 (0.37)

52. Secondary Outcome: Change From Baseline in the Wechsler Intelligence Scale for Children - Fourth Edition (WISC-IV) Digit Span Subtotal Scores at Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 51
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 24
units on a scale
  Digit Span Forward: Scaled Process Score | 0.53 (0.50)
  Digit Span Backward: Scaled Process Score | 0.36 (0.52)

53. Secondary Outcome: Number of Participants With a Response (Response Rate) up to Week 8
Description: Response rate analysis compared the frequency of response between LY2216684 treatment groups versus placebo for participants who had a final study period II (weeks 1-8) Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHD-RS-IV-PV:IR) total score <=60% of their baseline total score. ADHD-RS-IV-PV:IR measures 18 symptoms in Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) ADHD diagnosis. Item scores range: 0 (none/never or rarely) to 3 (severe/very often). Total scores range: 0 to 54.
Time Frame: Baseline, up to 8 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Placebo | LY2216684 (0.1 mg/kg/Day) | LY2216684 (0.2 mg/kg/Day) | LY2216684 (0.3 mg/kg/Day)
Number analyzed (Participants) | 63 | 58 | 60 | 59
Participants | 22 | 19 | 34 | 28

54. Secondary Outcome: Number of Participants With a Response (Response Rate) up to Week 8 in Stimulant Naive Methylphenidate Group
Description: as for outcome 53
Time Frame: Baseline, up to 8 weeks
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Methylphenidate
Number analyzed (Participants) | 26
Participants | 14

ADVERSE EVENTS:
Groups:
- Placebo - Treatment Phase: Participants were given the placebo in both tablet (LY2216684 placebo) and capsule (methylphenidate placebo) forms QD po for the 8-week double-blind treatment phase.
- LY2216684 (0.1 mg/kg/Day) - Treatment Phase: Participants were given 0.1 milligrams per kilogram per day (mg/kg/day) of LY2216684 in tablet form QD po for the 8-week double-blind treatment phase. Participants were also given placebo capsules to maintain methylphenidate blinding.
- LY2216684 (0.2 mg/kg/Day) - Treatment Phase: Participants were given 0.2 mg/kg/day of LY2216684 in tablet form QD po for the 8-week double-blind treatment phase. Participants were also given placebo capsules to maintain methylphenidate blinding.
- LY2216684 (0.3 mg/kg/Day) - Treatment Phase: Participants were given 0.3 mg/kg/day of LY2216684 in tablet form QD po for the 8-week double-blind treatment phase. Participants were also given placebo capsules to maintain methylphenidate blinding.
- Methylphenidate - Treatment Phase: Participants were given 18 mg/day to 54 mg/day of extended-release methylphenidate capsules, based on weight QD po for the 8-week double-blind treatment phase. Participants were also given placebo tablets to maintain LY2216684 blinding.
- Placebo - Taper Phase: Methylphenidate blind: Participants were given the placebo in capsule form QD po for the 2-week taper phase.
- LY2216684 (0.1 mg/kg/Day) - Taper Phase; LY2216684 (0.3 mg/kg/Day) - Taper Phase: Participants were given the reduced dose of LY2216684 in tablet form QD po for 2 weeks of tapering in the taper phase.
- LY2216684 (0.2 mg/kg/Day) - Taper Phase: Participants were given the reduced dose of LY2216684 in tablet form QD po for 2 weeks of tapering in taper phase.
- Methylphenidate - Taper Phase: Participants were given the placebo in capsule form QD po for the 2-week taper phase.
Arm/Group | Placebo - Treatment Phase | LY2216684 (0.1 mg/kg/Day) - Treatment Phase | LY2216684 (0.2 mg/kg/Day) - Treatment Phase | LY2216684 (0.3 mg/kg/Day) - Treatment Phase | Methylphenidate - Treatment Phase | Placebo - Taper Phase | LY2216684 (0.1 mg/kg/Day) - Taper Phase | LY2216684 (0.2 mg/kg/Day) - Taper Phase | LY2216684 (0.3 mg/kg/Day) - Taper Phase | Methylphenidate - Taper Phase
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/76 | 0/75 | 0/75 | 0/36 | 0/10 | 0/15 | 0/7 | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 51/78 | 58/76 | 59/75 | 49/75 | 30/36 | 1/10 | 4/15 | 0/7 | 0/12 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Phase (N=78) | LY2216684 (0.1 mg/kg/Day) - Treatment Phase (N=76) | LY2216684 (0.2 mg/kg/Day) - Treatment Phase (N=75) | LY2216684 (0.3 mg/kg/Day) - Treatment Phase (N=75) | Methylphenidate - Treatment Phase (N=36) | Placebo - Taper Phase (N=10) | LY2216684 (0.1 mg/kg/Day) - Taper Phase (N=15) | LY2216684 (0.2 mg/kg/Day) - Taper Phase (N=7) | LY2216684 (0.3 mg/kg/Day) - Taper Phase (N=12) | Methylphenidate - Taper Phase (N=4)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8) | 14 (16) | 3 (3) | 11 (16) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (6) | 13 (18) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (8) | 9 (10) | 10 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 4 (4) | 10 (10) | 7 (7) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 7 (8) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 6 (6) | 10 (10) | 8 (9) | 17 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 4 (6) | 6 (7) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (16) | 11 (13) | 14 (16) | 9 (16) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 4 (4) | 7 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 4 (6) | 14 (15) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 2 (3) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (5) | 4 (4) | 2 (2) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Some sites may have received data with identifying information from the central lab; data from 69 participants were excluded from efficacy analyses. Data were excluded from efficacy analyses for a participant randomized before study site approval.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days